CLINICAL TRIAL: NCT05139641
Title: Multidisciplinary Shared Decision Making of Fertility Preservation in Young Women With Breast Cancer
Acronym: MYBC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MedicalExcellence (Other)
Collaborators: Asan Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MYBC
Record Dates: First submitted 2021-11-17; First posted 2021-12-01 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Young Womenwith Breast Cancer

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control group (Placebo Comparator)
  Interventions: Behavioral: Counseling to preserve fertility
- counseling theraphy (Experimental)
  Interventions: Behavioral: Counseling to preserve fertility
- Retrospective data (No Intervention)

INTERVENTIONS:
Behavioral: Counseling to preserve fertility — Counseling to preserve fertility VS Control group
  Arms: control group; counseling theraphy

SUMMARY:
Multidisciplinary shared decision making of fertility preservation in Young womenwith Breast Cancer (MYBC): A Pragmatic stepped wedge cluster randomised trial

ELIGIBILITY:
Inclusion Criteria:

* Women aged 19 to 40 years old
* A person diagnosed with breast cancer by biopsy
* Those who don't have evidence of distant metastasis
* Eastern Cooperative Oncology Group(ECOG) performance status: 0-2 score
* Before registering for clinical trials, chemotherapy, radiation therapy, anti-hormone therapy, immunotherapy, and surgery are not performed
* A person who has fully understood and listened to the explanation of this clinical trial and then gave written consent

Exclusion Criteria:

* Histologically, a person diagnosed with follicular or sarcoma
* Those with a history of breast cancer (including recurrent breast cancer)
* A person diagnosed with another cancer before breast cancer
* A person diagnosed with metastatic breast cancer
* A person who has a mental illness and has a hard time understanding clinical trials
* Those who plan to conduct follow-up observation elsewhere(to change of hometowm)
* Menopausal factors without menstruation after more than a year from the last menstrual date
* A pregnant woman
* Inappropriate for participation in clinical trials

Ages: 19 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4100 (Estimated)
Dates: Start 2021-12 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
selection ratio of fertility preservation procedure | selection ratio of fertility preservation procedure from Baseline to six years

SECONDARY OUTCOMES:
The success rate of pregnancy | The success rate of pregnancy from Baseline to six years

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Excellence, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Baek SY, Kim HK, Park S, Yu JH, Lee MH, Youn HJ, Kim HA, Han JH, Choi JE, Lee JR, Lee KH, Chung S, Chae HD, Kim S, Yoo S, Hahm SK, Kim HJ. Multidisciplinary Shared Decision Making for Fertility Preservation in Young Women With Breast Cancer. J Breast Cancer. 2023 Dec;26(6):582-592. doi: 10.4048/jbc.2023.26.e44. Epub 2023 Oct 11. PMID 37985382